CLINICAL TRIAL: NCT07326566
Title: A Phase 2 Randomized, Multicenter Study to Evaluate the Efficacy and Safety of Silevertinib, an Oral EGFR Inhibitor, in Combination With Temozolomide in Patients With Newly Diagnosed Glioblastoma With Unmethylated MGMT Promoter and EGFRvIII
Brief Title: Study of Silevertinib With Temozolomide for the Treatment of Newly Diagnosed GBM With Unmethylated MGMT and EGFRvIII
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Black Diamond Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BDTX-1535-201
Record Dates: First submitted 2026-01-07; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma (GBM); Newly Diagnosed Glioblastoma; GBM; Glioblastoma Multiforme (GBM); Glioma; Central Nervous System Diseases; Brain Cancer
Keywords: EGFR; Glioblastoma; Unmethylated; Unmethylated MGMT promoter; Newly Diagnosed; temozolomide; Temodar; silevertinib; BDTX-1535; EGFR alterations; epidermal growth factor receptor; EGFRvIII; epidermal growth factor receptor (EGFR)
MeSH Terms: conditions — Glioblastoma; Glioma; Central Nervous System Diseases; Brain Neoplasms | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- silevertinib and temozolomide (Experimental): silevertinib at dose determined in Part 1 until disease progression in combination with temozolomide 150-200 mg/m2 orally once daily on Days 1 to 5 of each 28-day cycle for maximum of 6 cycles
  Interventions: Drug: silevertinib in combination with temozolomide
- temozolomide (Active Comparator): temozolomide 150-200 mg/m2 orally once daily on Days 1 to 5 of each 28-day cycle for maximum of 6 cycles
  Interventions: Drug: temozolomide (TMZ)

INTERVENTIONS:
Drug: silevertinib in combination with temozolomide — Participants enrolled into Part 1 (Safety Lead-In) or randomized to Arm A in Part 2 will receive silevertinib at dose determined in Part 1 until disease progression in combination with temozolomide 150-200 mg/m2 orally once daily on Days 1 to 5 of each 28-day cycle for maximum of 6 cycles.
  Other Names: BDTX-1535; Temodar; TMZ
  Arms: silevertinib and temozolomide
Drug: temozolomide (TMZ) — Participants randomized to Arm B will receive temozolomide 150-200 mg/m2 orally once daily on Days 1 to 5 of each 28-day cycle for maximum of 6 cycles
  Other Names: TMZ; Temodar
  Arms: temozolomide

SUMMARY:
The purpose of this study is to see if combining silevertinib with temozolomide after surgery and radiotherapy helps treat newly diagnosed glioblastoma (GBM) better than using temozolomide alone in the maintenance setting.

Specifically, this study is being done to find answers to the following questions:

* How much of the study drugs (silevertinib combined with temozolomide) should be given to participants with GBM?
* What are the side effects participants have when taking the study drug (silevertinib combined with temozolomide)?
* Can the study drug (silevertinib combined with temozolomide) help participants with GBM live longer without disease progression compared to treatment with temozolomide alone?

DETAILED DESCRIPTION:
Silevertinib was designed to block a growth signal important to some cancers where tumors grow because of changes in a protein called epidermal growth factor receptor (EGFR). These changes are called gene amplifications, mutations, or alterations and are found in tumors. Temozolomide is a drug that fights cancer cells by damaging DNA (the genetic material of cells), which could cause the tumor cells to die. It is the standard treatment for adults with certain types of newly diagnosed brain cancer, like GBM. It is given together with radiotherapy and sometimes afterward as maintenance therapy.

This study has 2 parts. To be eligible for the study, participants must have received a diagnosis of GBM, had surgery to remove or reduce the size of the tumor, and received adjuvant radiation therapy and temozolomide. No other prior treatments for GBM are allowed.

In Part 1 (called the Safety Lead-in), participants will receive silevertinib combined with temozolomide to determine if the combination is safe and to find the best dose. Approximately 12 participants are expected to enroll in Part 1 of the study.

In Part 2, all participants will be randomized to one of two different treatment groups:

* Group 1: Silevertinib + temozolomide
* Group 2: Temozolomide only

Approximately 150 participants are expected to be randomized in Part 2 of the study.

In both Part 1 and Part 2, the study treatment will be given in "cycles". Each cycle will be 28 days. After a cycle ends, the next cycle will immediately begin the next day. Both silevertinib and temozolomide will be taken orally. Silevertinib is taken daily until disease progression and temozolomide is taken for the first 5 days of each cycle (up to 6 cycles).

If participants are found to be eligible for the study and enrolled (in Part 1) or randomized (in Part 2), participants will:

* Take the study drug as directed
* Return for frequent clinic visits to monitor overall health and status of GBM
* Undergo imaging and other laboratory tests to determine status of GBM
* Complete a paper diary at home to record the date and time(s) that the study drug is taken

ELIGIBILITY:
Key Inclusion Criteria:

* Newly diagnosed histologically confirmed glioblastoma that is isocitrate dehydrogenase wild type (IDH-WT).
* Positive EGFR status in the brain tumor as determined by a commercially available test or validated laboratory assay (CLIA or comparable certification).
* For Part 1 (Safety Lead-in) ONLY: EGFR alterations.
* For Part 2 (Randomized, Controlled Trial) ONLY: EGFRvIII.
* For Part 2 (Randomized, Controlled Trial) ONLY: Unmethylated MGMT promoter tumor status based on a validated assay.
* No treatment for newly diagnosed GBM other than surgery followed by standard-of-care adjuvant postoperative radiation (54 to 60 Gy) and TMZ chemotherapy.
* At least 4 weeks since completion of radiation therapy, with a post-radiation MRI showing no progression.

Key Exclusion Criteria:

* Recurrent multifocal disease, metastatic, leptomeningeal, or extracranial GBM, or gliomatosis cerebri.
* Progression of GBM prior to Enrollment, Screening, or Randomization.
* Biopsy-only/no resectional surgery.
* Prior or concomitant treatment for GBM with an EGFR-targeting agent, including silevertinib, bevacizumab, cytotoxic chemotherapy, immunotherapy, experimental therapies, Gliadel wafers, GammaTile®, or other intratumoral or intracavitary antineoplastic therapy.
* Intent to use Optune® (TTF).
* Significant other uncontrolled health conditions or other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) | 12 months
  Progression-free survival, defined as the time from the date of randomization to the date of first disease progression per RANO 2.0 by BICR assessment or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival | 18 months
  Overall survival defined as time from first dose of study drug to death from any cause.

IPD SHARING:
Plan to Share IPD: No